CLINICAL TRIAL: NCT06313359
Title: Fall Risk and Quality of Life: Influence of Dual Task Performance, Cognition, and Sensorimotor Variables in Individuals With Cancer Treatment Related Peripheral Neuropathy.
Brief Title: Fall Risk and Quality of Life: in Individuals With Cancer Treatment Related Peripheral Neuropathy.
Status: Recruiting | Type: Observational
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Priya Karakkattil, Assistant Professor, Texas Woman's University
Other Study IDs: FY2024-125
Record Dates: First submitted 2024-03-01; First posted 2024-03-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cancer treatment induced peripheral neuropathy: Individuals with a history of non CNS cancer with cancer treatment induced peripheral neuropathy symptoms.
- Control group: Age and gender matched individuals without peripheral neuropathy symptoms.

SUMMARY:
The purpose of this research is to examine the impact of peripheral neuropathy on fall risk and quality of life in people who had cancer and neuropathy from cancer treatments. The investigators are interested to find out if the participant have any difficulty with thinking, feeling, balancing, or moving around that will contribute to risk for falls or quality of life. Investigators are also interested to see if the participants have any difficulty with doing two activities at the same time, such as walking and texting.

DETAILED DESCRIPTION:
Cancer related cognitive impairment (CRCI) is a common side effect of treatment of cancer during and after chemotherapy and is seen in patients with non-central nervous system( non-CNS) cancer. Though common after chemotherapy, other treatments such as hormone therapies and targeted therapies can also cause cognitive deficits.. The self-reported prevalence of cognitive complains in cancer survivors was 75% in a large web based study with non CNS cancers . The clinical presentation of these cognitive impairments include memory deficits, difficulty with learning attention, concentration, reasoning, processing speed, executive functions and visuospatial skills. Therefore the cognitive impairment can have a negative impact on quality of life, daily functioning and ability to work in patients with cancer while undergoing treatment and while in remission.

Acquired Peripheral Neuropathy (APN) is another common side effect of treatment for cancer. While majority of the peripheral neuropathy symptoms are due to neurotoxic chemotherapy agents resulting in chemotherapy-induced peripheral neuropathy (CIPN), neuropathy symptoms can also occur as paraneoplastic, immune-mediated, or neoplastic neuropathies. The reported prevalence of CIPN is 68% within first month after chemotherapy and continued to be present in 47% of the survivors even 6 years later. The clinical presentation of the CIPN includes numbness, tingling, or burning, neuropathic pain, decrease of muscle tone and coordination, and loss of balance. The symptoms tends to begin distally in the fingers and toes and moves proximally through the extremities. CIPN is typically associated with treatment using platinum based drugs, taxanes, epothilones, vinca alkaloids, bortezomib and thalidomide.

Individuals with CIPN are significantly more likely to suffer falls and fall related injuries. In breast cancer survivors with neuropathy, 40.9% experienced falls on both flat surfaces and non-flat surfaces during upright activities. Gait is a complex functional activity that requires the integration of the musculoskeletal, sensory, neurological, and cognitive systems. Significant gait variability in step width and step length with forward walking has been reported in cancer survivors with peripheral neuropathy compared to healthy controls. However, normal daily walking does not include just walking in a forward direction, but rather it involves walking in different directions such as walking backwards to sit in a chair. Although gait variability has been reported with forward walking, the gait variability while walking backwards in patients with cancer with APN has not been investigated previously.

Cognitive impairment has been strongly associated with decreased performance in dual task abilities and higher number of falls in older adults. Performing concurrent tasks such as walking and talking or walking and texting is a normal aspect of life. Concurrent performance of two tasks with distinct motor and cognitive demands has been associated with increased fall risk in older adults. Ability to do such dual task (DT) has shown to be declined in persons with cognitive and motor impairments. Ability to perform DT has been also reported to be affected in persons with diabetic peripheral neuropathy. There is only one reported study that evaluated the cognitive and sensory deficits associated with orbital stability in gait on treadmill during single and dual task in cancer survivors with and without peripheral neuropathy. However, walking on the treadmill at fixed speed does not translate to the real-world adaptations on overground walking in different directions with the added challenge of a cognitive task. Though cognitive and peripheral neuropathy symptoms are reported in patients with non- CNS cancers who are undergoing treatment and while in remission, ability to perform dual task with forward and backward walking has not been assessed in this population and not compared with an age and gender matched control without peripheral neuropathy. Additionally, it is important to investigate what cognitive, motor and sensory impairments can predict fall risk and decreased quality of life in this population compared to an age and gender matched control.

The purpose of this proposed exploratory pilot study is to evaluate the dual task cost of variable walking in individuals diagnosed with cancer treatment induced peripheral neuropathy compared to age and gender matched individuals without peripheral neuropathy. backward walking on an over ground computerized mat. A secondary purpose will be to identify what type of cognitive, motor and sensory impairments can correlate quality of life in individuals diagnosed with cancer treatment induced peripheral neuropathy and can predict fall risk in this population compared to compared to age and gender.

ELIGIBILITY:
Inclusion Criteria:

Experimental group

* Individuals 18 years and older
* diagnosed with non- CNS cancer who underwent treatment and presents with peripheral neuropathy symptoms.

Control group

* age (+/- one year) and gender matched individuals
* no diagnosed peripheral neuropathy
* No diagnosed cognitive symptoms.

Exclusion Criteria:

* Unable to follow two step commands.
* Unable to ambulate x 50 feet independently without use of an assistive device.
* Unable to use a phone to send text messages.
* Diagnosis of diabetic peripheral neuropathy
* Diagnosis of CNS cancer.
* Unable to speak/understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non CNS Cancer population with neuropathy symptoms related to cancer treatments.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Fall risk | 5 minutes
  Fall risk will be assessed using the Timed Up and Go (TUG)-Test. For the TUG, the participant will be asked to stand up from a chair, walk 3 m and touch a line on the floor, walk back to the chair and sit down. Timing of the test will begin when the tester gives the command "go" and will be stopped when the participant made contact with the chair as they sat down.
Quality of life- in cancer patients | 5 minutes
  Participants in the cancer related peripheral neuropathy group will complete the Functional Assessment of Cancer Therapy- General (FACT-G ) to assess self-reported quality of life. The FACT-G uses a 5-point Likert scale, with higher numbers indicating a better health state.

SECONDARY OUTCOMES:
Trail Making Test (TMT) Parts A & B | 5 minutes
  Trail Making Test assesses attention, psychomotor, and higher-level cognitive function and has been recommended to be used to in cancer population. The time it takes to complete the parts A and B will be recorded in seconds
Single Task- Working Memory | 3 minutes
  Single task assessment of working memory will be assessed by randomly picking one of the following tests (serial sevens (7s), spelling words backwards or recite months backwards) for 30 seconds in seated position.
Single Task- Visual Attention Cognitive Task | 3 minutes
  Visual-attention cognitive tasks will be tested by randomly selecting one of the following texting activity for 30 seconds (texting animal names, cities, or colors on a smart phone) in a seated position.
Protective Sensation | 5 minutes
  Protective sensation in the upper and lower extremities will be measured using the Semmes-Weinstein monofilament.
Grip Strength | 5 minutes
  Grip strength will be assessed using a Jamar handheld dynamometer.
LE strength assessment- HHD | 10 minutes
  Muscle strength testing of the ankle dorsiflexors, knee flexors, knee extensors, hip flexors, hip extensors and hip abductors using a handheld dynamometer using a make test.
Dynamic Balance | 5 minutes
  Dynamic balance and coordination will be assessed using the Four-Square Step Test (FSST).
Single Task- Gait Speed | 8 minutes
  For the single task gait component, we will utilize the Zeno© Electronic Walkway for assessing walking in both forward and backward directions using self-selected speed. Participants will commence/continue walking two feet prior to and after contacting the electronic walkway to account for acceleration and deceleration.
Dual Task- Working Memory & Gait Speed - Composite measure | 5 minutes
  Participants will complete three trials of walking forward and three trials of walking backward with simultaneous execution of a randomly selected working memory task (serial sevens (7s), spelling words backwards or recite months backwards)
Dual Task- Visual Attention Cognitive Task & Gait Speed - Composite measure | 5 minutes
  Participants will complete three trials of walking forward and three trials of walking backward with simultaneous execution of a randomly selected visual-attention cognitive task (texting animal names, cities, or colors on a smart phone)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Karakkattil, PhD, Principal Investigator — Texas Woman's University; Asha Vas, PhD, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Staff NP, Grisold A, Grisold W, Windebank AJ. Chemotherapy-induced peripheral neuropathy: A current review. Ann Neurol. 2017 Jun;81(6):772-781. doi: 10.1002/ana.24951. Epub 2017 Jun 5. PMID 28486769
- [Background] Small GH, Brough LG, Neptune RR. The influence of cognitive load on balance control during steady-state walking. J Biomech. 2021 Jun 9;122:110466. doi: 10.1016/j.jbiomech.2021.110466. Epub 2021 Apr 23. PMID 33962328
- [Background] Mounier NM, Abdel-Maged AE, Wahdan SA, Gad AM, Azab SS. Chemotherapy-induced cognitive impairment (CICI): An overview of etiology and pathogenesis. Life Sci. 2020 Oct 1;258:118071. doi: 10.1016/j.lfs.2020.118071. Epub 2020 Jul 14. PMID 32673664
- [Background] Montero-Odasso M, Sarquis-Adamson Y, Kamkar N, Pieruccini-Faria F, Bray N, Cullen S, Mahon J, Titus J, Camicioli R, Borrie MJ, Bherer L, Speechley M. Dual-task gait speed assessments with an electronic walkway and a stopwatch in older adults. A reliability study. Exp Gerontol. 2020 Dec;142:111102. doi: 10.1016/j.exger.2020.111102. Epub 2020 Oct 2. PMID 33017671
- [Background] Lange M, Joly F, Vardy J, Ahles T, Dubois M, Tron L, Winocur G, De Ruiter MB, Castel H. Cancer-related cognitive impairment: an update on state of the art, detection, and management strategies in cancer survivors. Ann Oncol. 2019 Dec 1;30(12):1925-1940. doi: 10.1093/annonc/mdz410. PMID 31617564
- [Background] Komatsu H, Yagasaki K, Komatsu Y, Yamauchi H, Yamauchi T, Shimokawa T, Doorenbos AZ. Falls and Functional Impairments in Breast Cancer Patients with Chemotherapy-Induced Peripheral Neuropathy. Asia Pac J Oncol Nurs. 2019 Jul-Sep;6(3):253-260. doi: 10.4103/apjon.apjon_7_19. PMID 31259221
- [Background] Autissier E. Chemotherapy-Induced Peripheral Neuropathy: Association With Increased Risk of Falls and Injuries. Clin J Oncol Nurs. 2019 Aug 1;23(4):405-410. doi: 10.1188/19.CJON.405-410. PMID 31322611